CLINICAL TRIAL: NCT02538796
Title: The Embodied Cognition: Exploratory Study of Automatic and Controlled Processes in Anorexia Nervosa. A Monocentric Study
Brief Title: The Embodied Cognition: Exploratory Study of Automatic and Controlled Processes in Anorexia Nervosa.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1001179; 2010-A01523-36 (Other: ANSM)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Cognition; Conscious; Non-Conscious
MeSH Terms: conditions — Anorexia Nervosa | interventions — Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Patients group 1 (Experimental): TEA + Grober Test + Task 1 + Grober Test
  Interventions: Other: TEA + Grober Test + Task 1 + Grober Test
- Patients group 2 (Experimental): TEA + Grober Test + Task 2 + Grober Test
  Interventions: Other: TEA + Grober Test + Task 2 + Grober Test
- Patients group 3 (Experimental): TEA + Grober Test + Implicit Task 3 + Grober Test
  Interventions: Other: TEA + Grober Test + Implicit Task 3 + Grober Test
- Patients group 4 (Experimental): TEA + Grober Test + Explicit Task 3 + Grober Test
  Interventions: Other: TEA + Grober Test + Explicit Task 3 + Grober Test
- Healthy volonteers group 1 (Active Comparator): TEA + Grober Test + Task 1 + Grober Test
  Interventions: Other: TEA + Grober Test + Task 1 + Grober Test
- Healthy volonteers group 2 (Active Comparator): TEA + Grober Test + Task 2 + Grober Test
  Interventions: Other: TEA + Grober Test + Task 2 + Grober Test
- Healthy volonteers group 3 (Active Comparator): TEA + Grober Test + Implicit Task 3 + Grober Test
  Interventions: Other: TEA + Grober Test + Implicit Task 3 + Grober Test
- Healthy volonteers group 4 (Active Comparator): TEA + Grober Test + Explicit Task 3 + Grober Test
  Interventions: Other: TEA + Grober Test + Explicit Task 3 + Grober Test

INTERVENTIONS:
Other: TEA + Grober Test + Task 1 + Grober Test — The Test of Everyday Attention (TEA) measures the reaction time of the participant during the occurrence of an expected stimulus.
  The Grober Test with 16 words to learn and to remember, measures the episodic verbal memory long term.
  The Task 1 consists of a stimulus that moves on the screen. The response of the patient is done on the keyboard. It is composed on two conditions: one is fast (without conscious), the other consists in assessing words (conscious). It includes food and non-food words.
  Arms: Healthy volonteers group 1; Patients group 1
Other: TEA + Grober Test + Task 2 + Grober Test — The TEA measures the reaction time of the participant during the occurrence of an expected stimulus.
  The Grober Test with 16 words to learn and to remember, measures the episodic verbal memory long term.
  The Task 2 consists of a stimulus that is fixed on the screen. The response of the patient is done by pushing or pulling a lever. It is composed on two conditions: one is fast (without conscious), the other consists in assessing words (conscious). It includes food and non-food words.
  Arms: Healthy volonteers group 2; Patients group 2
Other: TEA + Grober Test + Implicit Task 3 + Grober Test — The TEA measures the reaction time of the participant during the occurrence of an expected stimulus.
  The Grober Test with 16 words to learn and to remember, measures the episodic verbal memory long term.
  The Task 3 is a compilation of tasks 1 and 2 to investigate the bidirectional link. The instructions are implicit condition to detect an A in the word ("yes-no" answer).
  Arms: Healthy volonteers group 3; Patients group 3
Other: TEA + Grober Test + Explicit Task 3 + Grober Test — The TEA measures the reaction time of the participant during the occurrence of an expected stimulus.
  The Grober Test with 16 words to learn and to remember, measures the episodic verbal memory long term.
  The Task 3 is a compilation of tasks 1 and 2 to investigate the bidirectional link. The instructions are explicit condition to judge the emotional value of words ("positive-negative" answer).
  Arms: Healthy volonteers group 4; Patients group 4

SUMMARY:
Anorexia nervosa (AN) is a common psychiatric illness, with severe prognosis (5% mortality) that has changed little over in half a century. One of the forms is the restrictive anorexia nervosa (ANR). It consists of a phobia of weight gain and food with a massive food restriction. This pathology is studied in psychology but not using the theories of embodied cognition in which "perception and action" interact through sensorimotor processes. They are the source of attitudes (unconscious) towards certain stimuli and influence our interpretation (conscious).

DETAILED DESCRIPTION:
The investigators hypothesis is that food restriction behavior is the result of two processes. One automatic and not conscious, which is an attraction toward food and manifests itself in the motivational attitudes of approach, and the other controlled and conscious, which prevents attraction to this type of stimuli and is manifested by motivational attitudes avoidance. These processes of attraction and avoidance are observed in embodied cognition paradigms because the answers induce movement of approach or avoidance of stimuli. The validation of these assumptions could lead to reconsideration of the respective roles of automatic and controlled processes in food behaviors of anorexics patients and to complete or refocus psychological techniques of care.

ELIGIBILITY:
Inclusion Criteria for patients:

* Restrictive anorexia nervosa according to Diagnostic and Statistical Manual of Mental Disorders Text Revision (DSM IV-TR)
* BMI> 16 to avoid the effects of undernutrition
* Start disorders <10 years
* Right handed
* Having given free and informed consent prior to study participation
* Subject affiliated to the French National Health Insurance

Inclusion Criteria for control group:

* BMI between 18,5 and 25
* Right handed
* Of school level paired in that of the patients (+/-1 the year)
* Having given free and informed consent prior to study participation
* Subject affiliated to the French National Health Insurance

Exclusion Criteria for patients and control group:

* Patients with at the beginning or during the study form of purgative anorexia nervosa
* Control with disorders of current or past eating behavior.
* Control making a restrictive diet during the study period
* Participants with depressive table
* Participants with a somatic problem restricted movement or a problem of uncorrected visual acuity annoying reading of the screen.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Response time (ms) in the different conditions of the three tasks (composite measure) | Day 1
  Tasks are:
  * tap a key on the computer keyboard during the presentation of food and non-food words containing an "A" on a computer screen
  * pull a lever towards you at the presentation of food and non-food words on a computer screen
  * pull a lever towards you at the presentation of food and non-food words that approach on a computer screen

SECONDARY OUTCOMES:
BMI in kg/m² | Day 1
  The Body Mass Index (BMI) is defined as the body mass divided by the square of the body height.
Rate of wrong answers | Day 1
  It is the rate of wrong answers in the different conditions of the three tasks.
Score EDI-2 | Day 1
  The Eating Disorder Inventory (EDI) is a self-report questionnaire used to assess the presence of eating disorders.
Silhouettes test score | Day 1
  The patient selects among several silhouettes a silhouette to represent her real body image and her ideal body image.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MASSOUBRE, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France